CLINICAL TRIAL: NCT01392495
Title: An Open-label Extension Study to CQTI571A2102 to Evaluate the Long-term Safety, Tolerability and Efficacy of QTI571 (Imatinib) in the Treatment of Severe Pulmonary Arterial Hypertension
Brief Title: Extension to CQTI571A2102 to Evaluate Long-term Safety, Tolerability and Efficacy of Imatinib in Severe Pulmonary Arterial Hypertension (PAH)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Novartis discontinued the development of imatinib in PAH due to requirement of regulatory authorities for additional data to secure marketing approval in PAH.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CQTI571A2102E1; 2010-021960-14 (EudraCT Number)
Record Dates: First submitted 2011-07-11; First posted 2011-07-12 (Estimated); Results first posted 2015-07-13 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-07

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary arterial hypertension; imatinib; 6MWD
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- QTI571 (Experimental): Participants received 200 mg or 400 mg every day (qd) based on their highest tolerated dose in CQTI571A2102 (NCT01392469).
  Interventions: Drug: Imatinib

INTERVENTIONS:
Drug: Imatinib — 200 mg or 400 mg qd

SUMMARY:
This study was an extension to study CQTI571A2102 and was to evaluate the long-term safety, tolerability and efficacy of QTI571 (imatinib) in severe pulmonary arterial hypertension patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who completed in CQTI571A2102 clinical trial including all Study Completion assessments at the end of study visit met the eligibility criteria for that study and did not meet withdrawal criteria for safety reasons during study conduct

Exclusion Criteria:

* Patients with left ventricular ejection fraction (LVEF) < 45%
* Patients with thrombocytopenia, platelet count < 50 x109/L (50 x 103/µL).
* Patients with uncontrolled systemic arterial hypertension, systolic pressure > 160 mmHg or diastolic pressure > 90 mmHg.
* Patients with a QTcF > 450 ms for males and > 470 ms for females in the absence of right bundle branch block.

Other protocol-defined inclusion/exclusion criteria may apply

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-06; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- Novartis Investigative Site, Mineola, New York, United States
- Novartis Investigative Site, Darlinghurst, New South Wales, Australia
- Novartis Investigative Site, Leuven, Belgium
- Novartis Investigative Site, Hanover, Germany
- Novartis Investigative Site, Roma, RM, Italy
- Novartis Investigative Site, Vilnius, Lithuania
- Novartis Investigative Site, London, United Kingdom

REFERENCES:
- [Derived] Frost AE, Barst RJ, Hoeper MM, Chang HJ, Frantz RP, Fukumoto Y, Galie N, Hassoun PM, Klose H, Matsubara H, Morrell NW, Peacock AJ, Pfeifer M, Simonneau G, Tapson VF, Torres F, Dario Vizza C, Lawrence D, Yang W, Felser JM, Quinn DA, Ghofrani HA. Long-term safety and efficacy of imatinib in pulmonary arterial hypertension. J Heart Lung Transplant. 2015 Nov;34(11):1366-75. doi: 10.1016/j.healun.2015.05.025. Epub 2015 Jun 11. PMID 26210752
- [Derived] Hoeper MM, Barst RJ, Bourge RC, Feldman J, Frost AE, Galie N, Gomez-Sanchez MA, Grimminger F, Grunig E, Hassoun PM, Morrell NW, Peacock AJ, Satoh T, Simonneau G, Tapson VF, Torres F, Lawrence D, Quinn DA, Ghofrani HA. Imatinib mesylate as add-on therapy for pulmonary arterial hypertension: results of the randomized IMPRES study. Circulation. 2013 Mar 12;127(10):1128-38. doi: 10.1161/CIRCULATIONAHA.112.000765. Epub 2013 Feb 12. PMID 23403476

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | QTI571
Started | 17
Received 200 mg | 4
Received 400 mg | 13
Completed | 1
Not Completed | 16
Not completed — Death | 3
Not completed — Administrative problems | 8
Not completed — Withdrawal by Subject | 2
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Groups:
- QTI571: Participants received 200 mg or 400 mg qd based on their highest tolerated dose in CQTI571A2102.
Arm/Group | QTI571
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.5 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events, Serious Adverse Events and Deaths
Description: Adverse event monitoring was conducted throughout the trial.
Time Frame: 144 weeks
Population: Safety Analysis Set: The safety analysis set included all participants who received at least one dose of study drug during the extension and had at least one post-baseline safety assessment.
Measure: Number; unit: Participants
Groups:
- QTI571 200 mg; QTI571 400 mg: Participants received 200 mg or 400 mg qd based on their highest tolerated dose in CQTI571A2102.
Arm/Group | QTI571 200 mg | QTI571 400 mg
Number analyzed (Participants) | 4 | 13
Participants
  Adverse Events (serious and non-serious) | 4 | 13
  Serious Adverse Events | 4 | 5
  Deaths | 2 | 1

2. Secondary Outcome: Change From Baseline in the Six Minute Walk Distance (6MWD)
Time Frame: baseline, 144 weeks
Population: The study terminated early. No statistical analysis was performed on the efficacy outcomes.
Arm/Group | QTI571 200 mg | QTI571 400 mg
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Time to Clinical Worsening (TTCW) Endpoints
Time Frame: 144 weeks
Population: The study terminated early. No statistical analysis was performed on the efficacy outcomes.
Arm/Group | QTI571 200 mg | QTI571 400 mg
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Medical Resource Utilization
Time Frame: 144 weeks
Population: The study terminated early. No statistical analysis was performed on the efficacy outcomes.
Arm/Group | QTI571 200 mg | QTI571 400 mg
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- QTI571 200mg; QTI571 400mg: Participants received 200 mg or 400 mg qd based on their highest tolerated dose in CQTI571A2102.
Arm/Group | QTI571 200mg | QTI571 400mg
Serious Adverse Events (participants affected / at risk) | 4/4 | 5/13
Other Adverse Events (participants affected / at risk) | 4/4 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QTI571 200mg (N=4) | QTI571 400mg (N=13)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Right ventricular failure (Cardiac disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Mesenteric panniculitis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Salivary gland cyst (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Catatonia (Psychiatric disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 1
Urethral haemorrhage (Renal and urinary disorders) | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QTI571 200mg (N=4) | QTI571 400mg (N=13)
Anaemia (Blood and lymphatic system disorders) | 2 | 3
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 1
Periorbital oedema (Eye disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 6
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 3
Toothache (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 4
Oedema peripheral (General disorders) | 1 | 3
Pyrexia (General disorders) | 0 | 2
Bacteriuria (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Ear infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 2
Haemophilus infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 6
Otitis externa (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Staphylococcal skin infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 3
Blood creatinine increased (Investigations) | 1 | 1
Blood potassium decreased (Investigations) | 0 | 2
Blood sodium decreased (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Scleroderma (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 2
Sleep disorder (Psychiatric disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.